CLINICAL TRIAL: NCT05966974
Title: Study of Elective AGN1 LOEP in Osteopenic and Osteoporotic Subjects - a Retrospective Analysis
Brief Title: GRACE - Study of AGN1 LOEP in Osteopenic and Osteoporotic Patients
Status: Completed | Type: Observational
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AGN-CIP-302
Record Dates: First submitted 2022-12-16; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis
Keywords: Bone mineral density; Femoral strength; Hip fracture; Local osteo-enhancement procedure; LOEP; Proximal femur
MeSH Terms: conditions — Osteoporosis; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with AGN1 LOEP

SUMMARY:
The study is designed as a retrospective, single-center study for subjects previously treated with the AGN1 LOEP Kit. This will be a non-randomized and non-blinded study. The study will collect retrospective data on the safety and performance of AGN1 LOEP of all subjects treated outside of any other clinical study protocols between September 2019 and November 2022. A prospective questionnaire will be included to evaluate self-reported subject experiences.

ELIGIBILITY:
Inclusion Criteria:

* Subject has previously received AGN1 LOEP treatment between September 2019 and November 2022.
* Subject has willingness to participate in the study.
* Subject can give written informed consent to allow for data collection.

Exclusion Criteria:

* The subject's AGN1 LOEP treatment was previously performed as part of a prior protocoled clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteopenic and osteoporotic subjects receiving AGN1 LOEP treatment of the proximal femur.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Subject satisfaction | Through study completion, an average of 1.1 years
  Satisfaction level of subjects as measured by a Visual Analog Scale. The scale ranges from the lowest possible satisfaction to the highest possible satisfaction.
Subject Safety | During the procedure
  Incidence of all adverse events and serious adverse events occurring intraoperative determined to be at least possibly related to the procedure and/or device.
Subject Safety | Through study completion, an average of 1.1 years
  Incidence of all adverse events and serious adverse events occurring post-AGN1 LOEP determined to be at least possibly related to the procedure and/or device.

CONTACTS AND LOCATIONS:
Locations (1):
- Vitaz, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No